CLINICAL TRIAL: NCT00721799
Title: F-18 Fluorothymidine (FLT) PET Imaging for Early Evaluation of Response to Chemoradiation Therapy in Patients With Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: F-18 Fluorothymidine PET Imaging for Early Evaluation of Response to Therapy in Head & Neck Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Yusuf Menda, Associate Professor, Radiology-Nuclear Medicine, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 200801758; 1R21CA130281 (NIH)
Record Dates: First submitted 2008-06-10; First posted 2008-07-24 (Estimated); Results first posted 2017-10-03 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Mouth Neoplasms; Oropharyngeal Neoplasms; Laryngeal Neoplasms; Head and Neck Neoplasms
Keywords: Positron-Emission Tomography; radiation therapy; cisplatin; chemotherapy; FLT
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms; Laryngeal Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FLT PET scan (Experimental): Subjects receive 2 18F-Fluorothymidine PET scans
  * Scan 1 at baseline (within 30 days prior to the start of chemotherapy and radiation therapy)
  * Scan 2 between fraction 5 and 6 of radiation therapy (after 10 Gray of radiation)
  Interventions: Drug: 18F-Fluorothymidine PET scan

INTERVENTIONS:
Drug: 18F-Fluorothymidine PET scan — 18F-Fluorothymidine (0.04 - 0.08 mCi / kg to a maximum dose of 5 mCi) administered once intravenously for a positron emission tomography (PET) scan.
  Other Names: FLT; FLT PET scan

SUMMARY:
This is an imaging protocol only, not a therapeutic study.

The primary goal of the proposed study is to examine the utility of a new imaging study, Positron Emission Tomography with F-18 Fluorothymidine (FLT PET), in the early treatment evaluation of head and neck cancer. FLT uptake in the tumor correlates with the rate of cell proliferation. It is therefore hoped that changes in tumor FLT uptake after therapy will reflect change in the number of actively dividing tumor cells and will provide early assessment of treatment response.

Research subjects will undergo one PET scan with FLT. The scan is done prior to any therapeutic intervention (radiation or chemotherapy) can be obtained up to 30 days prior to the start of therapy. The uptake of FLT in the tumor will be analyzed to see if it can be used as a predictor of treatment efficacy and/or outcome.

There is an optional biopsy component to this study. Should the attending physicians (primarily the otolaryngologists) believe that the subject can safely undergo an outpatient biopsy, and the subject agrees, a biopsy is performed. The biopsy will be done within 30 days prior to treatment, similar to FLT PET scans. Tissue from the biopsy will be analyzed for markers of cellular proliferation and these markers will be correlated with the findings of FLT PET scan.

There will be a 2-year clinical follow-up to assess for treatment outcomes, local control, and overall survival.

DETAILED DESCRIPTION:
There are approximately 40,000 new cases of head and neck cancer each year in the United States. Approximately two thirds of these patients present with locally advanced disease with either large disease at the primary site and/or spread to regional lymph node levels. Treatment options include surgery, radiotherapy, and chemotherapy, usually applied in combination for advanced disease. Despite aggressive treatment, the 5-year survival for locally advanced disease remains poor (overall, approximately 50%). To increase the efficacy of locoregional therapy, different treatment maneuvers are used including increased radiation dose, concurrent use of chemotherapy and radiation therapy and high dose intra-arterial chemotherapy. Unfortunately, the increased intensity of combined treatment also leads to greater treatment related morbidity and mortality. It is currently difficult to predict who will benefit from intensive chemoradiotherapy and who would be most effectively treated with other combinations such as surgery and postoperative radiotherapy.

It is predictable that the most immediate signal of a successful antitumor therapeutic regime will be a decrease in cellular proliferation in the tumor. Therefore, a tracer, which is taken up into and retained in cells as a function of their proliferative activity, should provide rapid information as to the effectiveness of the treatment. FLT is an ideal tracer in this setting as its uptake is a function of thymidine kinase activity. Thymidine kinase activity is an established marker of cellular proliferation. FLT can be imaged with a PET scanner and the FLT uptake in the tumor can be reliably quantified. Preliminary studies including at our institution also confirm accumulation of FLT in untreated head and neck cancers. The objective of our study is to evaluate the utility of FLT PET imaging in predicting the outcome of treatment in terms of locoregional control and disease-free survival in patients (i.e., progression free survival) with head and neck cancer as well as overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a written informed consent document.
* Subject must have histologically confirmed squamous cell carcinoma of the head and neck.
* Subject must be scheduled to receive combined chemo-radiotherapy treatment for their standard cancer care. Treatment decisions will be made by the treating otolaryngologist, radiation, and medical oncologists.
* Male or females ≥ 18 years of age. Squamous cell cancer of the head and neck is exceedingly rare in children and not generally applicable to the pediatric population.
* Karnofsky greater than or equal to 60% at time of screening.
* Life expectancy of greater than 6 months.
* Subject must have normal organ and marrow function (as defined below) within 30 days of study enrollment:
* leukocytes ≥ 3,000/μL
* absolute neutrophil count ≥1,500/μL
* platelets ≥ 100,000/μL
* total bilirubin ≤ 1.0 mg/dl*
* Either AST OR ALT ≤ 2.5 X institutional upper limit of normal
* creatinine ≤ 1.5 x institutional upper limit of normal
* PT and PTT (if biopsy is to be performed) < 2.0 X upper normal limits
* The effects of FLT on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A screening urine hCG will be administered in the Nuclear Medicine to women of childbearing potential before each FLT scan and pregnant women will not be accepted as subjects in this study.

Exclusion Criteria:

* Subjects who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Subject may not be receiving any other investigational agents.
* Subject with a Karnofsky score of below 60.
* Pregnant women are excluded from this study. FLT PET has potential for teratogenic effects. Because there are potentially unknown risks for adverse events in nursing infants secondary to treatment of the mother with FLT, breastfeeding should be discontinued if the mother is imaged with FLT and may not resume for 48 hours after the FLT imaging.
* Subjects taking nucleoside analog medications such as those used as antiretroviral agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-03-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Menda, M.D., Principal Investigator — University of Iowa; John M. Buatti, M.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared through clinicaltrials.gov and in provision with the filed data sharing plan for the grant. Consent was not obtained from participants to share individual patient data.

REFERENCES:
- [Result] Menda Y, Boles Ponto LL, Dornfeld KJ, Tewson TJ, Watkins GL, Schultz MK, Sunderland JJ, Graham MM, Buatti JM. Kinetic analysis of 3'-deoxy-3'-(18)F-fluorothymidine ((18)F-FLT) in head and neck cancer patients before and early after initiation of chemoradiation therapy. J Nucl Med. 2009 Jul;50(7):1028-35. doi: 10.2967/jnumed.108.058495. Epub 2009 Jun 12. PMID 19525472
- [Result] Menda Y, Ponto LL, Dornfeld KJ, Tewson TJ, Watkins GL, Gupta AK, Anderson C, McGuire S, Schultz MK, Sunderland JJ, Graham MM, Buatti JM. Investigation of the pharmacokinetics of 3'-deoxy-3'-[18F]fluorothymidine uptake in the bone marrow before and early after initiation of chemoradiation therapy in head and neck cancer. Nucl Med Biol. 2010 May;37(4):433-8. doi: 10.1016/j.nucmedbio.2010.02.005. PMID 20447554
- [Result] Juweid ME, Thomas D, Menda Y, Tewson T, Graham MM, Herrmann K, Buck AK, Fayad L. PET/CT with 18F-FLT is unlikely to cause significant hepatorenal or hematologic toxicity. J Nucl Med. 2010 May;51(5):824-5. doi: 10.2967/jnumed.110.075945. No abstract available. PMID 20439512
- See also: The Holden Comprehensive Cancer Center — http://www.uihealthcare.com/depts/cancercenter/index.html

RESULTS

PARTICIPANT FLOW:
Groups:
- FLT PET: Subjects who receive F-18 Fluorothymidine [FLT]PET imaging prior to treatment.
  F-18 Fluorothymidine: FLT PET scan [0.04 to 0.08 mCi/kg (maximum of 5 mCi +/- 10%)]
Period: Overall Study
Arm/Group | FLT PET
Started | 33
Recieved FLT PET Scan 1 | 26
Received FLT PET Scan #2 | 25
Completed | 25
Not Completed | 8
Not completed — Withdrawal by Subject | 7
Not completed — withdraw by subject after scan 1 | 1

BASELINE CHARACTERISTICS:
Arm/Group | FLT PET
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Mean Pre-therapy FLT Uptake (SUVmean) in Predicting Progression Free Survival (PFS)
Description: Prediction efficacy is estimated using a hazard ratio (HR) and C-statistic (C-stat). Progression free survival is defined as the span of time from day 1 of therapy to date of disease recurrence (measured in months). Results are pooled with subjects from a pilot RDRC study for a total of 27 subjects analyzed.
Time Frame: 36 months
Population: Participants who underwent the pre-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: standardized uptake value (SUV)
Groups:
- FLT PET Scan: Subjects receive 2 18F-Fluorothymidine PET scans
  * Scan 1 at baseline (within 30 days prior to the start of chemotherapy and radiation therapy)
  * Scan 2 between fraction 5 and 6 of radiation therapy (after 10 Gray of radiation)
  F-18 Fluorothymidine dose = 0.04 to 0.08 mCi/kg (maximum of 5 mCi +/- 10%).
  Imaging technology: PET scan
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 27
standardized uptake value (SUV) | 4.23 (1.46)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.08, Regression, Cox; Hazard Ratio (HR) = 0.47
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.04, Regression, Cox; C-statistic = 0.73

2. Primary Outcome: Efficacy of Maximum Pre-therapy FLT Uptake (SUVmax) in Predicting Progression Free Survival (PFS)
Description: as for outcome 1
Time Frame: 36 months
Population: Participants who underwent the pre-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: standardized uptake value (SUV)
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 27
standardized uptake value (SUV) | 6.36 (2.21)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.05, Regression, Cox; Hazard Ratio (HR) = 0.42
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.02, Regression, Cox; C-statistic = 0.75

3. Primary Outcome: Efficacy of Pre-therapy Metabolic Tumor Volume in Predicting Progression Free Survival (PFS)
Description: Metabolic tumor volume using the FLT PET tracer. Prediction efficacy is estimated using a hazard ratio (HR) and C-statistic (C-stat). Progression free survival is defined as the span of time from day 1 of therapy to date of disease recurrence (measured in months). Results are pooled with subjects from a pilot RDRC study for a total of 27 subjects analyzed.
Time Frame: 36 months
Population: Participants who underwent the pre-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: mm^3 (cubic milimeters)
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 27
mm^3 (cubic milimeters) | 47.86 (32.49)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p < 0.01, Regression, Cox; Hazard Ratio (HR) = 2.44
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.02, Regression, Cox; C-statistic = 0.74

4. Primary Outcome: Efficacy of FLT Flux (K-FLT) Pre-therapy in Predicting Progression Free Survival (PFS)
Description: Prediction efficacy is estimated using a hazard ratio (HR) and C-statistic (C-stat). Progression free survival is defined as the span of time from day 1 of therapy to date of disease recurrence (measured in months). Results are pooled with subjects from a pilot RDRC study for a total of 27 subjects analyzed. FLT uptake in the tumor is a dynamic process that involves facilitated diffusion in and out of the cell and molecular changes in FLT. The rate, measured in mL/g/min, is a composite of the rate of transport of FLT from blood into the tissue and the transfer from tissue back into the blood, as well as the rate of molecular change of FLT.
Time Frame: 36 months
Population: Participants who underwent the pre-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: mL/g/min
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 27
mL/g/min | 0.07 (0.03)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.73, Regression, Cox; Hazard Ratio (HR) = 1.12
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.88, Regression, Cox; C-statistic = 0.52

5. Primary Outcome: Efficacy of the Patlak Influx Rate Constant for FLT (K-Patlak) Pre-therapy in Predicting Progression Free Survival (PFS)
Description: Prediction efficacy is estimated using a hazard ratio (HR) and C-statistic (C-stat). Progression free survival is defined as the span of time from day 1 of therapy to date of disease recurrence (measured in months). Results are pooled with subjects from a pilot RDRC study for a total of 27 subjects analyzed. The Patlak influx rate, measured in l /min, is the rate of transport of FLT from blood into the tissue as well as the rate of molecular change of FLT, using a Patlak analysis.
Time Frame: 36 months
Population: Participants who underwent the pre-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: l/min
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 27
l/min | 0.04 (0.02)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.78, Regression, Cox; Hazard Ratio (HR) = 1.11
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.66, Regression, Cox; C-statistic = 0.45

6. Primary Outcome: Efficacy of Pretherapy Total Lesion Proliferation in Predicting Progression Free Survival (PFS)
Description: as for outcome 1
Time Frame: 36 months
Population: Participants who underwent the pre-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: standardized uptake value (SUV)
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 27
standardized uptake value (SUV) | 143.68 (96.18)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.01, Regression, Cox; Hazard Ratio (HR) = 2.25
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.05, Regression, Cox; C-statistic = 0.70

7. Primary Outcome: Efficacy of Mean Mid-therapy FLT Uptake (SUVmean) in Predicting Progression Free Survival (PFS)
Description: Prediction efficacy is estimated using a hazard ratio (HR) and C-statistic (C-stat). Progression free survival is defined as the span of time from day 1 of therapy to date of disease recurrence (measured in months). Results are pooled with subjects from a pilot RDRC study for a total of 25 subjects analyzed.
Time Frame: 36 months
Population: Participants who underwent the mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: standardized uptake value (SUV)
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
standardized uptake value (SUV) | 2.53 (1.15)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.63, Regression, Cox; Hazard Ratio (HR) = 0.83
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.46, Regression, Cox; C-statistic = 0.58

8. Primary Outcome: Efficacy of Maximum Mid-therapy FLT Uptake (SUVmax) in Predicting Progression Free Survival (PFS)
Description: as for outcome 7
Time Frame: 36 months
Population: Participants who underwent the mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: standardized uptake value (SUV)
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
standardized uptake value (SUV) | 3.85 (1.80)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.58, Regression, Cox; Hazard Ratio (HR) = 0.81
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.36, Regression, Cox; C-statistic = 0.60

9. Primary Outcome: Efficacy of FLT Flux (K-FLT) Mid-therapy in Predicting Progression Free Survival (PFS)
Description: Prediction efficacy is estimated using a hazard ratio (HR) and C-statistic (C-stat). Progression free survival is defined as the span of time from day 1 of therapy to date of disease recurrence (measured in months). Results are pooled with subjects from a pilot RDRC study for a total of 25 subjects analyzed. FLT uptake in the tumor is a dynamic process that involves facilitated diffusion in and out of the cell and molecular changes in FLT. The rate, measured in mL/g/min, is a composite of the rate of transport of FLT from blood into the tissue and the transfer from tissue back into the blood, as well as the rate of molecular change of FLT.
Time Frame: 36 months
Population: Participants who underwent the mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: mL/g/min
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
mL/g/min | 0.04 (0.02)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.89, Regression, Cox; Hazard Ratio (HR) = 0.94
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.42, Regression, Cox; C-statistic = 0.59

10. Primary Outcome: Efficacy of the Patlak Influx Rate Constant for FLT (K-Patlak) Mid-therapy in Predicting Progression Free Survival (PFS)
Description: Prediction efficacy is estimated using a hazard ratio (HR) and C-statistic (C-stat). Progression free survival is defined as the span of time from day 1 of therapy to date of disease recurrence (measured in months). Results are pooled with subjects from a pilot RDRC study for a total of 25 subjects analyzed. The Patlak influx rate, measured in l /min, is the rate of transport of FLT from blood into the tissue as well as the rate of molecular change of FLT, using a Patlak analysis.
Time Frame: 36 months
Population: Participants who underwent the mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: l/min
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
l/min | 0.02 (0.02)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.43, Regression, Cox; Hazard Ratio (HR) = 1.29
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.80, Regression, Cox; C-statistic = 0.47

11. Primary Outcome: Efficacy of Mid-therapy Total Lesion Proliferation in Predicting Progression Free Survival (PFS)
Description: as for outcome 7
Time Frame: 36 months
Population: Participants who underwent the mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: standardized uptake value (SUV)
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
standardized uptake value (SUV) | 101.26 (76.91)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.01, Regression, Cox; Hazard Ratio (HR) = 2.01
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.07, Regression, Cox; C-statistic = 0.69

12. Primary Outcome: Efficacy of Percent Change in Mean FLT Uptake (SUVmean) Between Scan 1 & 2 in Predicting Progression Free Survival (PFS)
Description: as for outcome 7
Time Frame: 36 months
Population: Participants who underwent both the pre-therapy and mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: percentage change in SUVmean
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
percentage change in SUVmean | -0.39 (0.18)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.18, Regression, Cox; Hazard Ratio (HR) = 1.58
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.25, Regression, Cox; C-statistic = 0.63

13. Primary Outcome: Efficacy of Percent Change in Maximum FLT Uptake (SUVmax) Between Scans 1 & 2 in Predicting Progression Free Survival (PFS)
Description: as for outcome 7
Time Frame: 36 months
Population: Participants who underwent both the pre-therapy and mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: percentage change in SUVmax
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
percentage change in SUVmax | -0.39 (0.20)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.24, Regression, Cox; Hazard Ratio (HR) = 1.49
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.27, Regression, Cox; C-statistic = 0.62

14. Primary Outcome: Efficacy of Percent Change in FLT Flux (K-FLT) Between Scans 1 & 2 in Predicting Progression Free Survival (PFS)
Description: as for outcome 7
Time Frame: 36 months
Population: Participants who underwent both the pre-therapy and mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: percentage change in K-FLT
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
percentage change in K-FLT | -0.33 (0.21)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.99, Regression, Cox; Hazard Ratio (HR) = 1.00
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.84, Regression, Cox; C-statistic = 0.48

15. Primary Outcome: Efficacy of Percent Change the Patlak Influx Rate Constant for FLT (K-Patlak) Between Scans 1 & 2 in Predicting Progression Free Survival (PFS)
Description: as for outcome 7
Time Frame: 36 months
Population: Participants who underwent both the pre-therapy and mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: percentage change in K-Patlak
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
percentage change in K-Patlak | -0.51 (0.24)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.41, Regression, Cox; Hazard Ratio (HR) = 1.30
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.69, Regression, Cox; C-statistic = 0.54

16. Primary Outcome: Efficacy of Percent Change in the Total Lesion Proliferation Between Scans 1 & 2 in Predicting Progression Free Survival (PFS)
Description: as for outcome 7
Time Frame: 36 months
Population: Participants who underwent both the pre-therapy and mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
percentage change | -0.34 (0.14)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.17, Regression, Cox; Hazard Ratio (HR) = 1.56
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.18, Regression, Cox; C-statistic = 0.64

17. Primary Outcome: Efficacy of Mean Pre-therapy FLT Uptake (SUVmean) in Predicting Overall Survival (OS)
Description: Prediction efficacy is estimated using a hazard ratio (HR) and C-statistic (C-stat). Overall survival is defined as the span of time from day 1 of therapy to date of death from any cause (measured in months). Results are pooled with subjects from a pilot RDRC study for a total of 27 subjects analyzed.
Time Frame: 36 months
Population: Participants who underwent the pre-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: standardized uptake value (SUV)
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 27
standardized uptake value (SUV) | 4.23 (1.46)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.09, Regression, Cox; Hazard Ratio (HR) = 0.42
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.06, Regression, Cox; Hazard Ratio (HR) = 0.72

18. Primary Outcome: Efficacy of Maximum Pre-therapy FLT Uptake (SUVmax) in Predicting Overall Survival (OS)
Description: Prediction efficacy is estimated using a hazard ratio (HR) and C-statistic (C-stat). Progression free survival is defined as the span of time from day 1 of therapy to date of death from any cause (measured in months). Results are pooled with subjects from a pilot RDRC study for a total of 27 subjects analyzed.
Time Frame: 36 months
Population: Participants who underwent the pre-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: standardized uptake value (SUV)
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 27
standardized uptake value (SUV) | 6.36 (2.21)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.06, Regression, Cox; Hazard Ratio (HR) = 0.36
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.04, Regression, Cox; C-statistic = 0.74

19. Primary Outcome: Efficacy of Pre-therapy Metabolic Tumor Volume in Predicting Overall Survival (OS)
Description: Metabolic tumor volume using the FLT PET tracer. Prediction efficacy is estimated using a hazard ratio (HR) and C-statistic (C-stat). Overall survival is defined as the span of time from day 1 of therapy to date of death from any cause (measured in months). Results are pooled with subjects from a pilot RDRC study for a total of 27 subjects analyzed.
Time Frame: 36 months
Population: Participants who underwent the pre-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: mm^3 (cubic milimeters)
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 27
mm^3 (cubic milimeters) | 47.86 (32.49)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p < 0.01, Regression, Cox; Hazard Ratio (HR) = 3.01
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p < 0.01, Regression, Cox; C-statistic = 0.82

20. Primary Outcome: Efficacy of FLT Flux (K-FLT) Pre-therapy in Predicting Overall Survival (OS)
Description: Prediction efficacy is estimated using a hazard ratio (HR) and C-statistic (C-stat). Overall survival is defined as the span of time from day 1 of therapy to date of death from any cause (measured in months). Results are pooled with subjects from a pilot RDRC study for a total of 27 subjects analyzed. FLT uptake in the tumor is a dynamic process that involves facilitated diffusion in and out of the cell and molecular changes in FLT. The rate K-FLT, measured in mL/g/min, is a composite of the rate of transport of FLT from blood into the tissue and the transfer from tissue back into the blood, as well as the rate of molecular change of FLT.
Time Frame: 36 months
Population: Participants who underwent the pre-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: mL/g/min
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 27
mL/g/min | 0.07 (0.03)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.92, Regression, Cox; Hazard Ratio (HR) = 1.03
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.84, Regression, Cox; C-statistic = 0.48

21. Primary Outcome: Efficacy of the Patlak Influx Rate Constant for FLT (K-Patlak) Pre-therapy in Predicting Overall Survival (OS)
Description: Prediction efficacy is estimated using a hazard ratio (HR) and C-statistic (C-stat). Overall survival is defined as the span of time from day 1 of therapy to date of death from any cause (measured in months). Results are pooled with subjects from a pilot RDRC study for a total of 27 subjects analyzed. The Patlak influx rate, measured in l /min, is the rate of transport of FLT from blood into the tissue as well as the rate of molecular change of FLT, using a Patlak analysis.
Time Frame: 36 months
Population: Participants who underwent the pre-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: l/min
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 27
l/min | 0.4 (0.2)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.76, Regression, Cox; Hazard Ratio (HR) = 1.11
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.68, Regression, Cox; C-statistic = 0.45

22. Primary Outcome: Efficacy of Pretherapy Total Lesion Proliferation in Predicting Overall Survival (OS)
Description: as for outcome 17
Time Frame: 36 months
Population: Participants who underwent the pre-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: standardized uptake value (SUV)
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 27
standardized uptake value (SUV) | 143.68 (96.18)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p < 0.01, Regression, Cox; Hazard Ratio (HR) = 2.99
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.03, Regression, Cox; C-statistic = 0.74

23. Primary Outcome: Efficacy of Mean Mid-therapy FLT Uptake (SUVmean) in Predicting Overall Survival (OS)
Description: Prediction efficacy is estimated using a hazard ratio (HR) and C-statistic (C-stat). Overall survival is defined as the span of time from day 1 of therapy to date of death from any cause (measured in months). Results are pooled with subjects from a pilot RDRC study for a total of 25 subjects analyzed.
Time Frame: 36 months
Population: Participants who underwent the mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: standardized uptake value (SUV)
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
standardized uptake value (SUV) | 2.53 (1.15)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.55, Regression, Cox; Hazard Ratio (HR) = 0.78
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.35, Regression, Cox; C-statistic = 0.61

24. Primary Outcome: Efficacy of Maximum Mid-therapy FLT Uptake (SUVmax) in Predicting Overall Survival (OS)
Description: as for outcome 23
Time Frame: 36 months
Population: Participants who underwent the mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: standardized uptake value (SUV)
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
standardized uptake value (SUV) | 3.85 (1.80)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.48, Regression, Cox; Hazard Ratio (HR) = 0.74
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.28, Regression, Cox; C-statistic = 0.63

25. Primary Outcome: Efficacy of FLT Flux (K-FLT) Mid-therapy in Predicting Overall Survival (OS).
Description: Prediction efficacy is estimated using a hazard ratio (HR) and C-statistic (C-stat).Overall survival is defined as the span of time from day 1 of therapy to date of death from any cause (measured in months). Results are pooled with subjects from a pilot RDRC study for a total of 25 subjects analyzed. FLT uptake in the tumor is a dynamic process that involves facilitated diffusion in and out of the cell and molecular changes in FLT. The rate K-FLT, measured in mL/g/min, is a composite of the rate of transport of FLT from blood into the tissue and the transfer from tissue back into the blood, as well as the rate of molecular change of FLT.
Time Frame: 36 months
Population: Participants who underwent the mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: mL/g/min
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
mL/g/min | 0.04 (0.02)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.67, Regression, Cox; Hazard Ratio (HR) = 0.81
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.11, Regression, Cox; C-statistic = 0.71

26. Primary Outcome: Efficacy of the Patlak Influx Rate Constant for FLT (K-Patlak) Mid-therapy in Predicting Overall Survival (OS)
Description: Prediction efficacy is estimated using a hazard ratio (HR) and C-statistic (C-stat). Overall survival is defined as the span of time from day 1 of therapy to date of death from any cause (measured in months). Results are pooled with subjects from a pilot RDRC study for a total of 25 subjects analyzed. The Patlak influx rate, measured in l /min, is the rate of transport of FLT from blood into the tissue as well as the rate of molecular change of FLT, using a Patlak analysis.
Time Frame: 36 months
Population: Participants who underwent the mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: l/min
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
l/min | 0.02 (0.02)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.40, Regression, Cox; Hazard Ratio (HR) = 1.32
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.88, Regression, Cox; C-statistic = 0.48

27. Primary Outcome: Efficacy of Mid-therapy Total Lesion Proliferation in Predicting Overall Survival (OS)
Description: as for outcome 23
Time Frame: 36 months
Population: Participants who underwent the mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: standardized uptake value (SUV)
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
standardized uptake value (SUV) | 101.26 (76.91)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p < 0.01, Regression, Cox; Hazard Ratio (HR) = 2.39
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.03, Regression, Cox; C-statistic = 0.74

28. Primary Outcome: Efficacy of Percent Change in Mean FLT Uptake (SUVmean) in Predicting Overall Survival (OS)
Description: as for outcome 23
Time Frame: 36 months
Population: Participants who underwent both the pre-therapy and mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: percentage change in SUVmean
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
percentage change in SUVmean | -0.39 (0.18)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.26, Regression, Cox; Hazard Ratio (HR) = 1.51
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.46, Regression, Cox; C-statistic = 0.59

29. Primary Outcome: Efficacy of Percent Change in Maximum FLT Uptake (SUVmax) in Predicting Overall Survival (OS)
Description: as for outcome 23
Time Frame: 36 months
Population: Participants who underwent both the pre-therapy and mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: percentage change in SUVmax
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
percentage change in SUVmax | -0.39 (0.20)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.37, Regression, Cox; Hazard Ratio (HR) = 1.38
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.46, Regression, Cox; C-statistic = 0.59

30. Primary Outcome: Efficacy of Percent Change in FLT Flux (K-FLT) in Predicting Overall Survival (OS)
Description: as for outcome 23
Time Frame: 36 months
Population: Participants who underwent both the pre-therapy and mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: percentage change in K-FLT
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
percentage change in K-FLT | -0.33 (0.21)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.90, Regression, Cox; Hazard Ratio (HR) = 1.05
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.87, Regression, Cox; C-statistic = 0.52

31. Primary Outcome: Efficacy of Percent Change the Patlak Influx Rate Constant for FLT (K-Patlak) in Predicting Overall Survival (OS)
Description: as for outcome 23
Time Frame: 36 months
Population: Participants who underwent both the pre-therapy and mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: percentage change in K-Patlak
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
percentage change in K-Patlak | -0.51 (0.24)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.36, Regression, Cox; Hazard Ratio (HR) = 1.35
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.63, Regression, Cox; C-statistic = 0.56

32. Primary Outcome: Efficacy of Percent Change in the Total Lesion Proliferation in Predicting Overall Survival (OS)
Description: as for outcome 23
Time Frame: 36 months
Population: Participants who underwent both the pre-therapy and mid-therapy FLT PET scan
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FLT PET Scan
Number analyzed (Participants) | 25
percentage change | -0.34 (0.14)
Statistical Analysis 1: Comparison: FLT PET Scan; Test type: Other; p = 0.20, Regression, Cox; Hazard Ratio (HR) = 1.56
Statistical Analysis 2: Comparison: FLT PET Scan; Test type: Other; p = 0.24, Regression, Cox; C-statistic = 0.63

ADVERSE EVENTS:
Time Frame: 1 calendar day following injection with the tracer agent, FLT
Arm/Group | FLT PET
All-Cause Mortality (participants affected / at risk) | 6/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

LIMITATIONS AND CAVEATS:
* HPV (human papilloma virus) status of tumors not available.
* Therapy heterogeneity in the therapy; radiotherapy fairly consistent but chemotherapy regimens varied.
* Small sample size is limiting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes